CLINICAL TRIAL: NCT01133015
Title: Comparison of Fractional Flow Reserve and Minimal Luminal Area by Intravascular Ultrasound in Evaluating Intermediate Coronary Artery Stenosis in Each Coronary Artery
Brief Title: Comparison of Fractional Flow Reserve and Intravascular Ultrasound
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Keimyung University (Other); Inje University (Other); Ajou University (Other)
Responsible Party: Bon-Kwon Koo / Professor, Seoul National University hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1001-009-305
Record Dates: First submitted 2010-05-24; First posted 2010-05-28 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Stenosis
Keywords: FFR; IVUS; MLA
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intermediate lesion (Experimental): Intermediate lesion will be evaluated by both IVUS and FFR
  Interventions: Device: Fractional flow reserve; Device: IVUS

INTERVENTIONS:
Device: Fractional flow reserve — Fractional flow reserve measured by pressure wire
  Other Names: RADI pressure wire
Device: IVUS — intravascular ultrasound
  Other Names: Volcano IVUS, boston scientific

SUMMARY:
This study will evaluate the relationship of Fractional Flow Reserve (FFR) and Minimal Lumen Area (MLA) by IntraVascular UltraSound (IVUS) by comparing the results of the both tests which is done as a part of the cardiac catheterization.

DETAILED DESCRIPTION:
Invasive X-ray coronary angiography remains the "reference standard" for the evaluation of coronary artery stenoses. Recently, intravascular ultrasound (IVUS) has been introduced as an invasive method for the evaluation of coronary artery stenoses and has been shown to be highly accurate in stenosis detection when compared to X-ray angiography. While invasive X-ray angiography and IVUS evaluate morphological features of coronary arterial plaques, fractional flow reserve (FFR) is an invasive measure of the hemodynamic significance of a stenosis obtained in the catheterization laboratory by measuring changes in intracoronary arterial pressure before and after maximal vasodilation induced by intravenous adenosine. An FFR value less than 0.75 has been shown to predict ischemia in vascular beds distal to the stenosis by radionuclide perfusion modalities and has been shown to be associated with worse outcomes. Therefore, FFR is considered to be an invasive hemodynamic "reference standard" for the evaluation of the hemodynamic significance of coronary arterial stenoses. While IVUS can provide additional morphological information in intermediate stenoses, it can not provide further functional information.

We are currently conducting investigation in the validation of IVUS against FFR in intermediate coronary artery stenoses in each coronary arteries. However, the difference of the values of IVUS data in each coronary artery, eg. left anterior descending artery or right coronary artery, has not been validated against invasive hemodynamic measurements of fractional flow reserve in patients with intermediate stenoses by invasive X-ray angiography. We hypothesize that IVUS-derived measurements are interpreted differently in each coronary arteries in the diagnosis of hemodynamically significant coronary artery stenoses, using FFR as the reference standard in patients with coronary artery stenoses 40%< and <70%.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-85
* Presence of at least one obstructive coronary artery stenosis as defined by:
* Previous catheterization or CT angiogram with any lesion 70% or greater
* Previous positive functional stress test (this does not include CTA alone)
* Ability and Willingness to provide informed consent
* Ability and Willingness to perform required follow up procedures

Exclusion Criteria:

* History of coronary artery bypass graft surgery
* Previously revascularized lesion
* Creatinine>1.6 mg/dL or GFR<30 pre-procedure per institutional standards
* Known Pregnancy
* Inability to perform CTA
* Arrhythmia precluding diagnostic CT examination
* Contrast agent allergy that cannot be adequately premedicated
* Severe PVD precluding cardiac catheterization
* Patient not a candidate for IVUS and FFR
* Inability or unwillingness to provide informed consent
* Inability or unwillingness to perform required follow up procedures

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
lumen area | 1 day
  lumen area cut-off that can predict the functional significance of a lesion

SECONDARY OUTCOMES:
angiographic stenosis, % plaque area | 1 day
  angiographic and intravascular ultrasound parameters that can best predict the functional significance of lesions
CT measurement | 1 day
  Diagnostic accuracy of CT derived parameters

CONTACTS AND LOCATIONS:
Overall Officials: Bon-kwon Koo, MD/PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

REFERENCES:
- [Derived] Koo BK, Yang HM, Doh JH, Choe H, Lee SY, Yoon CH, Cho YK, Nam CW, Hur SH, Lim HS, Yoon MH, Park KW, Na SH, Youn TJ, Chung WY, Ma S, Park SK, Kim HS, Tahk SJ. Optimal intravascular ultrasound criteria and their accuracy for defining the functional significance of intermediate coronary stenoses of different locations. JACC Cardiovasc Interv. 2011 Jul;4(7):803-11. doi: 10.1016/j.jcin.2011.03.013. PMID 21777890